CLINICAL TRIAL: NCT00539968
Title: An Open-Label, Two-Part Study to Determine the Safety, Tolerability, and Activity of Lonafarnib and Docetaxel
Brief Title: A Study to Evaluate the Safety, Tolerability, and Activity of Lonafarnib and Docetaxel (Study P04467AM1)(TERMINATED)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P04467
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Prostate Cancer; Breast Cancer; Ovarian Cancer; Lung Cancer; Gastric Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Stomach Neoplasms | interventions — Docetaxel; lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel plus lonafarnib (single arm) (Experimental): Docetaxel plus lonafarnib
  Interventions: Drug: Docetaxel plus lonafarnib

INTERVENTIONS:
Drug: Docetaxel plus lonafarnib — Docetaxel: 60-75 mg/m2
  Lonafarnib: 150-375 mg PO BID
  Other Names: Docetaxel (Taxotere®); lonafarnib (SCH 066336, Sarasar®)

SUMMARY:
This study will determine the best doses of docetaxel and lonafarnib when the two anti-cancer agents are used in combination. Patients with tumors for which treatment with docetaxel would be appropriate are eligible. A second part of the study will further examine the effectiveness of the combination treatment in men with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1: Subjects may be male or female and must be at least 18 years of age.
* For Part 1: Cancer for which docetaxel treatment is appropriate.
* For Part 1: Docetaxel-naïve
* For Part 2: Subjects must be male and at least 18 years of age.
* For Part 2: Subjects must have adenocarcinoma of the prostate confirmed by histologic/cytologic biopsy.
* For Part 2: Subjects must have progressive, metastatic, AIPC and a PSA of 10 ng/ml or more after hormonal therapy prior to docetaxel treatment. Progressive disease is defined as a consistently increasing serum PSA level within 28 days prior to docetaxel administration.
* Adequate organ function within 3 weeks prior to first study drug administration.
* Performance status (ECOG) is less than or equal to 2.
* Subject understands and agrees to procedures and participation by signing informed consent form.
* Agrees to use medically accepted form of contraception.

Exclusion Criteria:

* Receipt of or need to continue to receive prohibited medications (listed in the protocol) more recently than the washout period (indicated in the protocol).
* Surgery within 3 weeks prior to first study drug administration.
* History within 5 years prior to first study drug administration of another malignancy except adequately treated Stage I/II basal/squamous cell skin cancer.
* Radiation therapy to more than 25% of his/her total bone marrow during life.
* Radiation therapy within 3 weeks prior to first study drug administration.
* Known hypersensitivity to prednisone, docetaxel, polysorbate 80, lonafarnib, or any excipients associated with these medications.
* Known contraindication to steroid use.
* Known leptomeningeal or CNS metastasis.
* Heart, vascular, or seizure disorder (detailed list in the protocol) within 6 months prior to first study drug administration.
* Baseline QTc interval greater than 450 msec.
* Grade 2 or more peripheral neuropathy or drug-related toxicity per CTCAE. Exceptions are noted in the protocol.
* Any clinically significant condition or situation that the investigator thinks would interfere with the study evaluations or subject's participation.
* Subject is part of staff personnel involved in the study.
* Subject has known clinically significant immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and dose-limiting toxicities | Until disease progression, unacceptable dose delays or reductions, or unacceptable toxicity
Rate of prostate-specific antigen (PSA) responses | Until disease progression, unacceptable dose delays or reductions, or unacceptable toxicity

SECONDARY OUTCOMES:
Proportion of subjects with dose-limiting toxicities | Until disease progression, unacceptable dose delays or reductions, or unacceptable toxicity
Plasma lonafarnib concentrations | Until disease progression, unacceptable dose delays or reductions, or unacceptable toxicity
RECIST-defined radiological response rate | Until disease progression, unacceptable dose delays or reductions, or unacceptable toxicity